CLINICAL TRIAL: NCT03538093
Title: Clinical and Functional Differences Between Local, Global and Mixed Lumbar Stabilization Exercises in Rehabilitation of Adult Patients With Lumbar Arthrodesis Surgery Due to Spinal Stenosis: a Randomized Clinical Trial
Brief Title: Lumbar Stabilization Exercises in Adult Patients With Lumbar Arthrodesis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Rodrigo Torres, Clinical Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCHILEKINEIT
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Arthrosis; Spine; Spinal Stenosis Lumbar
Keywords: arthrodesis; core stabilization; physical therapy
MeSH Terms: conditions — Osteoarthritis; Ankylosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Local Stabilization Exercise (Experimental): Experimental: Local Stabilization Exercise Consists of a standard inpatient and outpatient rehabilitation program which includes exercises that focuses the activation of the muscles considered as local stabilizers of the core (Transversus Abdominis and Multifidus).
  Interventions: Other: Experimental: Local Stabilization Exercise
- Global Stabilization Exercise (Experimental): Experimental: Global Stabilization Exercise Consists of a standard inpatient and outpatient rehabilitation program which includes exercises that focuses the activation of the muscles considered as global stabilizers of the core (Erector Spinae, Quadratus Lumborum, Abdominal External Oblique, Abdominal Internal Oblique and Rectus Abdominis).
  Interventions: Other: Experimental: Global Stabilization Exercise
- Mixed Stabilization Exercise (Experimental): Experimental: Mixed Stabilization Exercise Consists of a standard inpatient and outpatient rehabilitation program which includes exercises that focuses the activation of both local and global core stabilizer muscles.
  Interventions: Other: Experimental: Mixed Stabilization Exercise

INTERVENTIONS:
Other: Experimental: Local Stabilization Exercise — Inpatient phase (3-5 days): Day 1: lower limbs active mobilization on bed, abdominal breathing exercises, full body block twists. Day 2: manual transversus a. activation exercises, multifidus cross activation exercise, sitting on the edge of the bed. Day 3: bipedal stance, supervised gait reeducation, home care education, medical and physical therapy discharge with instructions.
  Outpatient phase:4th-6th week: hot compress + electrotherapy IFT (fr: 4kHz, AMF 100Hz, modulation 20Hz, 20 mins), stabilizer training. Hamstring, quadriceps, gluteus maximus and psoas stretching, stationary bicycle without load. 7th-9th week: stabilizer training elevating a leg, stationary bicycle low load. 10th-12th week: 1kg to elevated leg on stabilizer training, stationary bicycle moderate load.
  Arms: Local Stabilization Exercise
Other: Experimental: Global Stabilization Exercise — Inpatient phase (3-5 days): Day 1: lower limbs active mobilization on bed, abdominal breathing exercises, full body block twists. Day 2: add obliques cross exercises in supine with contralateral leg, lumbopelvic bridge exercises, sitting on the edge of the bed. Day 3: add bipedal stance, supervised gait reeducation, home care education, medical and physical therapy discharge with instructions.
  Outpatient phase: physiotherapy: 4th-6th week: hot compress + electrotherapy IFT, lumbopelvic bridge exercises, obliques cross exercises. Hamstring, quadriceps, gluteus maximus and medius stretching, stationary bicycle without load. 7th-9th week: FST, global exercises, stationary bicycle low load. 10th-12th week: physiotherapy, side plank, unilateral bridge, stationary bicycle moderate load.
  Arms: Global Stabilization Exercise
Other: Experimental: Mixed Stabilization Exercise — Inpatient phase (3-5 days): Day 1: lower limbs active mobilization on bed, abdominal breathing exercises, full body block twists. Day 2: manual transversus abdominis activation exercises, multifidus cross activation exercise, sitting on the edge of the bed. Day 3: bipedal stance, supervised gait reeducation, home care education, medical and physical therapy discharge with instructions.
  4th-6th week: hot compress + electrotherapy IFT, stabilizer training, hamstring, quadriceps, gluteus maximus and medius stretching, stationary bicycle without load. 7th-9th week: FST, global exercises, change stationary bicycle load to low load. 10th-12th week: physiotherapy, advanced global exercise (side plank), unilateral bridge,stationary bicycle moderate load.
  Arms: Mixed Stabilization Exercise

SUMMARY:
The purpose of this study is to determine which type of lumbar stabilization exercise is more effective to improve functionality and reduce pain in patients operated with lumbar arthrodesis, to guide clinical practice in the rehabilitation of these patients.

DETAILED DESCRIPTION:
The objective of this study is to determine which exercise modality (global, local or mixed) is most effective in reducing pain and improving function at 6 and 12 weeks after the operation. The methodology will be a randomized experimental clinical trial. The study population will be subjects who underwent surgery for lumbar spinal stenosis due to decompression and posterolateral fusion. The estimation of the sample size was made on the basis of the ANOVA test measures, following the guidelines established by Stevens, for which an α = 0.05 and β = 0.2 were used, power = 80% and moderate effect size. As a result, the program (GPower) gave us a total sample size of 24 subjects, so we will use a sample of 30 subjects due to the possibility of departure of some of them abandoning during the process. The sample will be taken from a waiting list of lumbar spinal stenosis surgery at the Traumatological Institute of Santiago (IT). To measure the level of functionality, we will use the Oswestry Disability Index 2.0 in Spanish, and for pain, the Visual Analogue Scale, in addition to recording general data. For each instrument, 3 measurements will be taken: preoperative, 6 and 12 weeks after the operation. To analyze the data, the program of the latest version of IBM SPSS Statistics Base will be used, a Shapiro Wilks normality test will be performed to confirm a normal distribution and then an ANOVA of repeated measures to confirm the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old, operated of lumbar spine arthrodesis for degenerative spinal stenosis at Traumatological Institute of Santiago de Chile

Exclusion Criteria:

* Overweight
* Underweight
* Previous Surgeries
* Postoperative complications
* Higher pain in lower limbs than in low back
* Inability to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Pain | 12 weeks
  Visual Analog Scale of pain. The range of the scale goes from 0 (no pain) to 10 (unbearable pain), and from a color spectrum between blue (0) and red (10). The result is measured as the distance (in milimeters), from 0 to the point the patient indicates.
Disability | 12 weeks
  Measured by Oswestry Disability Index, which ranges from 0 to 100. 0 is equated with no disability and 100 is the maximum disability possible.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Lecaros, MSc, Principal Investigator — Instituto Traumatológico Dr. Teodoro Gebauer Weisser
Locations (1):
- University of Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided